CLINICAL TRIAL: NCT04066517
Title: STereotactic RadioAblation by Multimodal Imaging for VT (STRA-MI-VT)
Acronym: STRA-MI-VT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Cardiologico Monzino (Other)
Collaborators: Istituto Europeo di Oncologia (Other)
Responsible Party: Principal Investigator, Corrado Carbucicchio, Head of Ventricular Intensive Care Unit, Centro Cardiologico Monzino
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R 918/19 - CCM968
Record Dates: First submitted 2019-07-24; First posted 2019-08-26 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Refractory Ventricular Tachycardia
MeSH Terms: conditions — Tachycardia, Ventricular

STUDY DESIGN:
Masking Description: No masking in this study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Open Label (Experimental): Non-randomized, open label clinical trial that intends to treat with SBRT 15 patients with refractory VT.
  Interventions: Procedure: SBRT

INTERVENTIONS:
Procedure: SBRT — Multimodal-imaging guided SBRT for VT ablation.

SUMMARY:
Study of multimodal-imaging guided stereotactic body radiotherapy (SBRT) for ventricular tachycardia (VT) ablation.

DETAILED DESCRIPTION:
STRA-MI-VT study is a spontaneous, open-label, not randomized, prospective clinical trial.

The objective of the study is to evaluate the safety and efficacy of SBRT in strictly selected patients with refractory VT.

Multimodal cardiac imaging combined with electroanatomic mapping to provide a specific patient's tailored SBRT treatment plan choosing amang different linear accelerators.

ELIGIBILITY:
Inclusion Criteria:

* ICD/S-ICD recipients with refractory VT
* Not eligible for conventional catheter ablation or -in alternative- that have undergone failing conventional catheter ablation attempts, refusing surgery for the treatment of the arrhythmia.
* LVEF ≥ 20%.
* Age ≥ 50 years.
* Signed an IRB approved written informed consent document.

Exclusion Criteria:

* Previous radiotherapy with cardiac involvement.
* Pregnancy or breastfeeding.
* Active myocardial ischemia.
* Acute revascularation in the past 120 days.
* Acute hemodynamic instability (cardiogenic shock/NYHA IV).
* Serious disease with presumed life expectancy less than 12 months.
* Any condition that is deemed a contraindication in the judgment of the investigators.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2025-06-13 (Estimated); Study Completion 2025-06-13 (Estimated)

PRIMARY OUTCOMES:
SBRT safety during 12 month follow-up | 12 months
  Serious adverse events will be defined using CTCAE v4.0 criteria.
SBRT efficacy based on reduction of VT episodes during 12 month follow-up | 12 months
  There will be 6 week blanking period after therapy to allow for ablation effect

SECONDARY OUTCOMES:
Total mortality | 12 months
Health related quality of life | 12 months
  Health related quality of life for positive or negative changes based on score from SF-36 Questionnaire
Cardiac functional changes | 12 months
  Cardiac functional changes evaluated by echocardiography ejection fraction

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Centro Cardiologico Monzino, IRCCS, Milan, MI
  - Istituto Europeo di Oncologia, IRCCS, Milan, MI

REFERENCES:
- [Background] Carbucicchio C, Jereczek-Fossa BA, Andreini D, Catto V, Piperno G, Conte E, Cattani F, Rondi E, Vigorito S, Piccolo C, Bonomi A, Gorini A, Pepa M, Mushtaq S, Fassini G, Moltrasio M, Tundo F, Marvaso G, Veglia F, Orecchia R, Tremoli E, Tondo C. STRA-MI-VT (STereotactic RadioAblation by Multimodal Imaging for Ventricular Tachycardia): rationale and design of an Italian experimental prospective study. J Interv Card Electrophysiol. 2021 Sep;61(3):583-593. doi: 10.1007/s10840-020-00855-2. Epub 2020 Aug 27. PMID 32851578
- [Background] Carbucicchio C, Andreini D, Piperno G, Catto V, Conte E, Cattani F, Bonomi A, Rondi E, Piccolo C, Vigorito S, Ferrari A, Pepa M, Giuliani M, Mushtaq S, Scara A, Calo L, Gorini A, Veglia F, Pontone G, Pepi M, Tremoli E, Orecchia R, Pompilio G, Tondo C, Jereczek-Fossa BA. Stereotactic radioablation for the treatment of ventricular tachycardia: preliminary data and insights from the STRA-MI-VT phase Ib/II study. J Interv Card Electrophysiol. 2021 Nov;62(2):427-439. doi: 10.1007/s10840-021-01060-5. Epub 2021 Oct 5. PMID 34609691